CLINICAL TRIAL: NCT02500355
Title: Carpal Tunnel Release With Partial Excision of the Flexor Retinaculum Through Two Small Incisions
Brief Title: Carpal Tunnel Release Via Two Small Incisions Comparing With Via Standard Incision And Under Endoscope
Acronym: CTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: qhd20150712
Record Dates: First submitted 2015-07-12; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Endoscopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Carpal Tunnel Release via limited approaches with 2 years follow-up.
  Interventions: Procedure: Carpal Tunnel Release via limited approaches
- Group B (Active Comparator): Carpal Tunnel Release via standard approach with 2 years follow-up.
  Interventions: Procedure: Carpal Tunnel Release via standard approach
- Group C (Placebo Comparator): Endoscopic Carpal Tunnel Release with 2 years follow-up.
  Interventions: Procedure: Endoscopic Carpal Tunnel Release; Device: endoscope or an arthroscopic device

INTERVENTIONS:
Procedure: Carpal Tunnel Release via limited approaches — Carpal tunnel release with partial excision of the flexor retinaculum via two small incisions.
  Arms: Group A
Procedure: Carpal Tunnel Release via standard approach — Carpal tunnel release with partial excision of the flexor retinaculum via the standard incision.
  Arms: Group B
Procedure: Endoscopic Carpal Tunnel Release — Carpal tunnel release under endoscope.
  Arms: Group C
Device: endoscope or an arthroscopic device
  Arms: Group C

SUMMARY:
Carpal Tunnel Release via Two Small Incisions Comparing With via Standard Incision And Under Endoscope.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) affects over 60 million people worldwide. If a regimen of conservative management has failed, surgical release of the median nerve is warranted. Numerous approaches for carpal tunnel release have been described that range from an open technique to a limited incision to endoscopic release. In addition, partial excision of the flexor retinaculum is advocated by some surgeons because of obtaining better outcomes. However, the procedure is difficult to be accomplished through small incisions owing to poor visualization. Currently, balance of incision, visualization, and partial excision of the flexor retinaculum is still controversial.

The objective of this report is to introduce carpal tunnel release with partial excision of the flexor retinaculum through two small incisions. The procedures were performed under lighted head magnifier. This is the first report on the use of our technique. For comparison, the investigators also included two other groups of standard open carpal tunnel release with partial excision of the flexor retinaculum and endoscopic carpal tunnel release without excision of the flexor retinaculum.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CTR was established based on Evidence for Surgical Treatment issued by the British Society for Surgery of the Hand (2003)
* Patients with moderate, severe, and very severe symptom.

Exclusion Criteria:

* Mild symptom.
* Finding had a ganglion based on preoperative ultrasound.
* Associated with infection, gout, or diabetes.
* Patients who discontinued intervention and lost to follow-up.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Severity of symptoms and functional status on Boston Questionnaire | 2 years

SECONDARY OUTCOMES:
Grip strength | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Study Chair — The Second Hospital of Qinhunangdao
Locations (1):
- The second hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Background] Notarnicola A, Maccagnano G, Tafuri S, Fiore A, Pesce V, Moretti B. Comparison of shock wave therapy and nutraceutical composed of Echinacea angustifolia, alpha lipoic acid, conjugated linoleic acid and quercetin (perinerv) in patients with carpal tunnel syndrome. Int J Immunopathol Pharmacol. 2015 Jun;28(2):256-62. doi: 10.1177/0394632015584501. Epub 2015 May 7. PMID 25953494
- [Result] Aksekili MA, Bicici V, Isik C, Aksekili H, Ugurlu M, Dogan M. Comparison of early postoperative period electrophysiological and clinical findings following carpal tunnel syndrome: is EMG necessary? Int J Clin Exp Med. 2015 Apr 15;8(4):6267-71. eCollection 2015. PMID 26131237